CLINICAL TRIAL: NCT02108314
Title: Physician-led Video-assisted Intervention for Increasing Mammography Uptake in Private Primary Care Practice in Singapore: A Cluster-Randomized Trial
Brief Title: Video-assisted Intervention for Increasing Mammography Uptake in Private Primary Care in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Dr Mark Chen, Assistant Professor, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 13-494
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Mammogram Scheduled
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Participants in the control arm were blinded as to the hypothesis of the study, undergoing a series of questions in about general health behaviours before their consultation, allowing the investigators to determine eligibility for the study. The associated participant information sheets for the control arm did not specifically mention breast cancer screening, maintaining blinding throughout. There was no reminder to the physician to promote mammography to participants. The physician continued with his or her usual counseling on health screening and mammography, if any. A 3-minute health promotion video by the Singapore Heart Foundation on healthy eating habits was administered to each participant, followed by a post-consultation questionnaire. The entire process took approximately 10 minutes.
- Video Screening and Counselling (Active Comparator): The intervention comprises 1) GP counseling, 2) 3-minute promotional video on mammography and 3) an informational brochure with relevant contact details and information for arranging a mammography screening. Pre- and post-consultation questionnaire were administered to participants to evaluate their health beliefs, with emphasis on breast cancer and mammography.
  Interventions: Behavioral: Video Screening and Counselling

INTERVENTIONS:
Behavioral: Video Screening and Counselling — The intervention comprises 1) GP counseling, 2) 3-minute promotional video on mammography and 3) an informational brochure with relevant contact details and information for arranging a mammography screening. Pre- and post-consultation questionnaire were administered to participants to evaluate their health beliefs, with emphasis on breast cancer and mammography.
  Arms: Video Screening and Counselling

SUMMARY:
Breast cancer is the leading female cancer in Singapore, but 3 in 5 women are not going for their regular mammography screenings at recommended frequencies despite 15 years of nationwide efforts by Breast Screen Singapore. The investigators aim to determine the efficacy of opportunistic health promotion for uptake of mammography screening in Singaporean women attending private sector primary care clinics in Singapore by implementing a simple and feasible questionnaire to identify potential candidates for mammography screening, coupled with recommendations by the primary care provider and a directed promotional video produced by Kandang Kerbau Hospital (KKH) that is aimed at addressing some of the barriers to screening.

DETAILED DESCRIPTION:
Breast cancer is the second leading cause of cancer-related deaths in women with an estimate of 508 000 deaths in 2011 worldwide . Incidence rates vary from 19.3 per 100,000 women in Eastern Africa to 89.7 per 100,000 women in Western Europe . Locally, 1 in every 16 Singaporean women in their lifetime is affected, making it the most common cancer in women in Singapore, with 17.9% of cancer deaths in women attributed to it. The Singapore Cancer Registry (2012) also revealed that the age-standardised incidence rates of newly diagnosed breast cancer have increased from 22.0 per 100,000 in the 1973-1977 period to 62.4 per 100,000 in the 2008-2012 period .

Studies have consistently shown that mammography is effective in early detection of breast cancer - , reducing breast cancer mortality of 20-22% . However, recent studies have questioned the efficacy of mammography. Gotszche et al. challenged that past trials had inadequate randomization , while a 1998 Cochrane Review questioned the potential confounding effect of advances in adjuvant chemotherapy (i.e. Tamoxifen) on overall breast cancer survival rates . With reference to the 2005 New England Journal of Medicine paper by Berry et al, screening remains an effective tool, and with therapy, has contributed to the decline in related mortality. In a 2011 local paper, Wang et al compared screen-detected and symptomatic women, concluding that screen-detected patients had an overall higher survival rates that their symptomatic counterparts .

For the past 15 years, the nationwide breast cancer-screening programme in Singapore has been recommending women aged 40-69 to undergo screening mammography, emphasizing that women in the younger age group of 40-49 should be screened once a year due to the unique local age-specific incidence rates showing an unusually high incidence of 34.4% in women aged 45-54 . Despite aggressive efforts and incentives, mammography uptake rates poor. A National Health Survey in 2010 revealed that 3 in 5 women are not going for their regular mammography at recommended frequencies . A pre-pilot study by Seow et al in 2009 showed that up to 27.4% of women surveyed had never had a mammogram before. A recent paper published in 2013 by Teo et al. also reported that regular mammography uptake rates are at a dismal rate of 26% . Dismal uptake rates are notably equally rampant in other countries, with a varying 40% to 90% of women quoted to be non-compliant to their respective breast cancer screening programmes . Local studies have revealed fear of pain and a belief that cancer would not happen to them as some barriers to screening . Teo et al. also revealed predictors of poor uptake as that of low income group, poor educational level, fear of pain/discomfort as well as being Malay. This illustrates the multidimensional influence of race, ethnicity, knowledge and health-seeking behavior in determining the compliance to regular screening.

With previous studies identifying various barriers to Singapore's mammography-screening program, the investigators hope to go further by evaluating the effectiveness of targeted interventions in helping women overcome said barriers. While there have been multiple trials done overseas - to determine the effectiveness of various interventions, there has only been two such local trials by Seow et al in 2012 and 1998 done in a public sector primary care setting - . As 80% of primary care in Singapore occurs in the private sector, conducting the study there would represent a different demographic of patient characteristics that has wider applicability. Furthermore, the strong doctor-patient relationship may help with the effectiveness of General Practitioner (GP)-based intervention. A key factor may therefore be lack of physician recommendation . Published evidence suggests patients were more likely to follow up with mammography screening when their primary care practitioner ordered testing - . As such, the investigators hope to design and evaluate a cost effective, feasible and relevant intervention that can be realistically implemented with the resources available in the workflow of the average GP clinic without additional resources and manpower requirements.

ELIGIBILITY:
Inclusion Criteria:

All women aged 40 - 69 years old registering at the clinic will be screened. For inclusion into either the intervention or control procedures, participants must be:

* Singapore citizens or Permanent Residents
* Women aged 40 - 69 years old who are not regularly undergoing mammography screening as per Singapore breast cancer screening guidelines, i.e.:

A) Not done a mammogram in the past 1 year if they are 40 to 49 years old B) Not done a mammogram in the past 2 years if they are 50 to 69 years old

Exclusion Criteria:

* Women who have already enrolled in the study (i.e. at a previous visit to the same or even other GP).
* Women who undergo regular mammography screenings (see above).
* Women with a personal history of breast cancer.
* Women who are unable to give informed consent (e.g. mentally incapacitated).
* Women who have requested to be excluded from the study.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mammography Uptake | 3 days after intervention
  The primary outcome is assessing the effectiveness of specific interventions in promoting mammography uptake in Singaporean females who are non-compliant to regular mammography. This was measured via self-reporting of mammography at 3 and 120 days.
Mammography Uptake | 120 days after intervention
  The primary outcome is assessing the effectiveness of specific interventions in promoting mammography uptake in Singaporean females who are non-compliant to regular mammography. This was measured via self-reporting of mammography at 3 and 120 days.

SECONDARY OUTCOMES:
Stages of behavior change | 3 days after intervention
  The investigators also measure if there is an intention to have a mammogram as indicated by making of an appointment, and intention to make an appointment based on self-reporting.
Stages of behavior change | 120 days after intervention
  The investigators also measure if there is an intention to have a mammogram as indicated by making of an appointment, and intention to make an appointment based on self-reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chen, PhD, Principal Investigator — NUHS; Fong Seng Lim, M.Med, Study Director — NUHS
Locations (1):
- Multiple General Practitioner Clinics in Singapore, Singapore, Singapore, Singapore